CLINICAL TRIAL: NCT05594030
Title: Thoracic Fluid Content by Electric Bioimpedance Versus Lung Ultrasound in Preterm Neonates With Respiratory Distress
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: MD 03/2022
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: preterm, respiratory distress, LUS, TFC
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Premature Birth; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective cohort study aims to evaluate the predictive value of thoracic fluid content measured by electric bioimpedance for detecting the need for surfactant administration or positive pressure ventilation requirement; whether invasive or non-invasive; in preterm neonates with respiratory distress and to compare it to lung ultrasound.

DETAILED DESCRIPTION:
Electrical cardiometry (bioimpedance) is an impedance-based method that has been recently introduced for continuous noninvasive hemodynamic monitoring for cardiac output (CO) and TFC in both term and preterm infants.

TFC is the sum of the total fluid volume found in the chest cavity; it is measured as the baseline resistance (bioimpedance) to the passage of a small electrical current through all chest tissues.

Larger TFC indicates a higher total thoracic fluid volume. TFC measurement has been correlated with heart failure symptoms, net fluid balance, and chest radiographic findings of abnormal pulmonary fluid content in adults.

Lung ultrasound (LUS) is a reliable technique for physicians to complement physical examination findings and has emerged as an alternative option to overcome the limitations of chest x rays (CXRs). Moreover, LUS shows better diagnostic accuracy than CXR in some critical conditions and has been successfully adapted in NICUs for the diagnosis of several diseases.

We thought that TFC monitoring may be able to predict the need for surfactant administration or positive pressure ventilation requirement; whether invasive or non-invasive; in preterm neonates with respiratory distress comparable to LUS.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates with gestational age ≤ 34 weeks, admitted with respiratory distress:

Defined as the presence of at least two of the following clinical symptoms:

Tachypnea, grunting, retractions (subcostal, intercostal, suprasternal), nasal flaring and other symptoms include apnea, bradypnea, irregular (seesaw) breathing, inspiratory stridor, wheezes and hypoxia

Exclusion Criteria:

* Preterm neonates with evidence of any of the following:

Chromosomal anomalies Mechanical ventilation or received endotracheal surfactant before first assessment

Ages: 1 Minute to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm neonates admitted to Ain shams University Hospital NICUs fulfilling the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
predictive value of thoracic fluid content measurement for detecting the need for surfactant administration or positive pressure ventilation requirement in preterm neonates with respiratory distress and to compare it to lung ultrasound. | 72 hours
  Thoracic fluid content will be measured on enrolment (TFC10 and follow up will be done after 3 days (TFC2) and at extubation from mechanical ventilation (TFC3) by electrical bioimpedance

SECONDARY OUTCOMES:
TFC parameters may offer the ability to monitor lung fluid content and provide longitudinal follow-up during interventions and disease processes. | 72 hours
  Thoracic fluid content will be measured on enrolment (TFC10 and follow up will be done after 3 days (TFC2) and at extubation from mechanical ventilation (TFC3) by electrical bioimpedance

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ain shams university, Cairo
  - Neonatal Intensive Care Units (NICUs), Ain Shams University, Cairo